CLINICAL TRIAL: NCT07022483
Title: A Phase 3, Multicenter, Randomized, Open-label Trial of Trastuzumab Deruxtecan Versus Standard of Care Chemotherapy With or Without Radiotherapy as Adjuvant Treatment for HER2-Expressing (IHC 3+/2+) Endometrial Cancer (DESTINY-Endometrial02/ GOG-3122/ ENGOT-en30/GINECO)
Brief Title: Study of Trastuzumab Deruxtecan Versus Standard of Care Chemotherapy for HER2-Expressing (IHC 3+/2+) Endometrial Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-854
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; cancer; T-DXd; HER2
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms | interventions — trastuzumab deruxtecan; Drug Therapy

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: T-DXd (Experimental): Participants will receive T-DXd 5.4 mg/kg intravenously (IV) once every 3 weeks (Q3W) with or without [optional] radiotherapy
  Interventions: Drug: Trastuzumab Deruxtecan
- Arm B: Standard of Care Chemotherapy (Active Comparator): Participants will receive carboplatin AUC 5 or 6 and paclitaxel 175 mg/m2 Q3W, or AUC 5 or 6 and paclitaxel 175 mg/m2 Q3W with or without [optional] radiotherapy or chemoradiotherapy (EBRT plus cisplatin [as radiosensitizer] 50 mg/m2
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — T-DXd will be administered at a dose of 5.4 mg/kg IV Q3W.
  Other Names: T-DXd; ENHERTU®
  Arms: Arm A: T-DXd
Drug: Chemotherapy — Carboplatin AUC 5 or 6 and paclitaxel will be administered at a dose of 175 mg/m2 Q3W, or carboplatin AUC 5 or 6 and paclitaxel 175 mg/m2 Q3W followed by chemoradiotherapy.
  Arms: Arm B: Standard of Care Chemotherapy

SUMMARY:
This study is designed to assess efficacy and safety of T-DXd adjuvant therapy, with or without radiotherapy, post-surgery in anticancer treatment naïve (including neoadjuvant therapy) endometrial cancer with various HER2 expression levels.

DETAILED DESCRIPTION:
This is a global, multicenter, open-label, phase 3 study to evaluate the efficacy and safety of T-DXd versus SoC chemotherapy with or without radiotherapy as adjuvant treatment in participants with HER2-expressing (IHC 3+/2+) endometrial cancer. Participants will be randomized 1:1 to either T-DXd or SoC chemotherapy. The primary objective will assess disease-free survival as assessed radiographically by BICR or by histopathologic confirmation of disease recurrence per local assessment.

T-DXd (Enhertu®) is a HER2 directed ADC composed of a humanized anti-HER2 IgG1 mAb with the same amino acid sequence as trastuzumab, which includes a plasma-stable, selectively cleavable linker and potent topoisomerase I inhibitor payload (a derivative of exatecan) that leverages the clinically validated DXd ADC technology.

ELIGIBILITY:
Key Inclusion Criteria

* Adults ≥18 years at the time the ICF is signed (Please follow local regulatory requirements if the legal age of consent for trial participation is >18 years old)
* Has histologically confirmed diagnosis of epithelial endometrial carcinoma. All histology's are allowed except for sarcomas (carcinosarcomas are allowed).
* Is newly diagnosed FIGO 2023 Stage IIC (including Stage IICmp53abn) or Stage III Note: FIGO 2023 Stage IIC includes disease with aggressive histological types (aggressive histological types are composed of high-grade EECs (grade 3), serous, clear cell, undifferentiated, mixed, mesonephric-like, gastrointestinal mucinous type carcinomas, and carcinosarcomas) with any myometrial involvement. FIGO 2023 Stage III includes disease with local and/or regional spread of the tumor of any histological subtype.
* Has HER2-expression (IHC 3+/2+) per 2016 ASCO-CAP gastric cancer IHC scoring guidelines as confirmed by central laboratory testing.
* Has adequate archived tumor tissue sample (sample from surgery is strongly recommended) available for assessment of HER2 status by central laboratory.

Key Exclusion Criteria

* Has uterine mesenchymal tumor such as an endometrial stromal sarcoma, leiomyosarcoma, or other types of pure sarcomas. Adenosarcomas are also not allowed.
* Has recurrent or FIGO 2023 Stage IV
* Has measurable residual tumor after surgery as determined by BICR assessment.
* Is known to have a POLE mutation from an approved and/or validated local test, according to local regulations, if available
* Has a medical history of MI within 6 months before randomization/enrollment, symptomatic CHF (NYHA Class II to IV). Participants with troponin levels above ULN at SCR (as defined by the manufacturer), and without any MI related symptoms should have a cardiologic consultation during SCR Period to rule out MI.
* Has a QTcF prolongation to > 480 msec based on average of the SCR triplicate12-lead ECG. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (ie, pulmonary emboli within 3 months of the trial enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion, etc.) and any autoimmune, connective tissue, or inflammatory disorder with potential pulmonary involvement (eg, rheumatoid arthritis, Sjogren's syndrome, sarcoidosis, etc.), or prior pneumonectomy.
* Has a history of (noninfectious) ILD/pneumonitis that required corticosteroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at SCR.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2032-03-23 (Estimated); Study Completion 2032-03-23 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival as Assessed by Blinded Independent Central Review or by Histopathologic Confirmation of Disease Recurrence per Local Assessment | From randomization to the first documented local regional recurrence, distant metastasis, or death due to any cause, whichever occurs first, up to approximately 51 months
  Disease-Free Survival will be assessed radiographically by BICR or by histopathologic confirmation of disease recurrence per local assessment.

SECONDARY OUTCOMES:
Overall Survival | From randomization to the date of death due to any cause, up to approximately 63 months
  Overall Survival is defined as the time interval from the date of randomization to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (40):
- United States (3):
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Trials365 LLC, Shreveport, Louisiana
  - Avera Medical Group Gynecologic Oncology Sioux Falls, Sioux Falls, South Dakota
- China (16):
  - Beijing Cancer Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Second University Hospital, Sichuan University, Chengdu
  - Obstetrics and Gynecology Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Cancer Hospital of Shandong First Medical University, Jinan
  - Linyi Cancer Hospital, Linyi
  - Jiangxi Maternal and Child Health Hospital, Nanchang
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning
  - Shanghai First Maternity and Infant HospitalShanghai First Maternity and Infant Hospital, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Yantai Yuhuangding Hospital, Yantai
- Japan (14):
  - Hyogo Cancer Center, Akashi-shi
  - NHO Kyushu Cancer Center, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Saitama Medical University International Medical Center, Hidaka-shi
  - Cancer Institute Hospital of JFCR, Kōtoku
  - Kurume University Hospital, Kurume-shi
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Gunma Prefectural Cancer Center, Ota-shi
  - NHO Hokkaido Cancer Center, Sapporo
  - Tohoku University Hospital, Sendai
  - Keio University Hospital, Shinjuku-ku
  - Mie University Hospital, Tsu
  - Yamagata University Hospital, Yamagata
- South Korea (3):
  - Keimyung University Dongsan Hospital, Daegu
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/